CLINICAL TRIAL: NCT07206095
Title: Integrative Diagnosis of Sickle Cell Disease (SCD) and Other Rare Anemia Disorders (RADs) for Personalized Medicine
Brief Title: Integrative Diagnosis for SCD and Other RADs
Acronym: INTEGRA
Status: Recruiting | Type: Observational
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Hospital Clinic de Barcelona, Barcelona, Spain (Unknown); Institute for Bioengineering of Catalonia (Other); Hospital Arnau de Vilanova, Lleida (Spain) (Unknown)
Responsible Party: Sponsor
Other Study IDs: PR(AMI)543/2020; Evidence 860436 (Other Grant/Funding Number: EC-H2020-MSCA-ITN-2019); Integra-SCD PI20/01454 (Other Grant/Funding Number: Instituto de Salud Carlos III (ISCIII)); GA 101095530 - SYNTHEMA (Other Grant/Funding Number: HORIZON-HLTH-2022-IND-13-02); GA 101017549 - GENOMED4ALL (Other Grant/Funding Number: H2020-SC1-FA-DTS-2020-1); PR(AMI)427/2021 (Other Grant/Funding Number: RADeep (Rare Anaemia Disorders European Epidemiological Platform))
Record Dates: First submitted 2025-09-16; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Sickle Cell Disease; Thalassaemia; Congenital Dyserythropoietic Anemia (CDA); Enzyme Disorder; Anemia; Spherocytosis, Hereditary; Stomatocytosis; Hemoglobin Disorder; Anemia Due to Membrane Defect; Rare Anemia Disorders
Keywords: SICKLE CELL DISEASE; RARE ANEMIA DISORDERS; PERSONALIZED MEDICINE; DIAGNOSIS; EKTACYTOMETRY
MeSH Terms: conditions — Anemia, Sickle Cell; Thalassemia; Anemia, Dyserythropoietic, Congenital; Anemia; Spherocytosis, Hereditary; Hemoglobinopathies; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: Analysis of genetic modifiers — Genetic modifiers for rare anemia disorders will be analyzed through massive sequencing.
Diagnostic Test: Disease phenotyping — Peripheral blood samples will be used for conventional phenotyping characterization including among others: RBCs morphology, fragility osmotic test, hemoglobin fraction and quantification, hemoglobin stability test, EMA binding test, RBC enzymes quantification assay, RBC rheological properties through Lorrca Maxsis Osmoscan/Oxygescan (Lorrca®)

SUMMARY:
INTEGRA aims at enabling personalized medicine for RHADs patients by the establishment of an integrative diagnostic approach based on deep phenotypic and genetic characterization through combining new generation methodologies.

DETAILED DESCRIPTION:
Objectives:

* To assess the prognostic value of LoRRca (ektacytometry) as biomarker providing information of SCD/RADs patients severity
* To investigate the correlation between LoRRca parameters and SCD/RADs patients genetic and phenotypic characterization.
* To identify genetic modifiers of RADs both new and previously described by GWAS as markers for prognosis and clinical course based on genomics approach.
* To establish an innovative algorithm for RADs patients characterization based on the integration of data generated through the analysis of genetic modifiers and the RBCs rheological properties by LoRRca profiles and microfluidics data in combination with RADs patients' clinical manifestations and treatments.
* To model the progression of RADs in a spleen-like filtering unit using microfluidic technologies to develop a novel diagnostic device for prognosis and patients' stratification. This device will be used for the characterization under flow of rheological and mechanical properties of single RBCs.
* To translate the results on a clinical practice recommendation for management of RADs patients endorsed by European Hematology bodies as ERN-EuroBloodNet and/or the European Hematology Association for its wide dissemination.

ELIGIBILITY:
Inclusion Criteria:

* Patients sustaining a confirmed or suspected diagnosis of an hereditary rare hemolytic anemia:
* Sickle cell disease
* Thalassemic syndromes
* Congenital dyserythropoietic anemia
* Enzymopathy
* Unstable Hemoblogin / Altered oxygen affinity
* Hereditary stomatocytosis
* Hereditary pyropoikilocytosis
* Hereditary spherocytosis with severe anemia (<8 g/dL) or inconclusive diagnosis:
* Patient with chronic hemolytic anemia and red cell smear compatible, but with:
* EMA binding test: inconclusive or negative
* Genetic testing: no definitive diagnosis (VUS or no findings)
* Not transplanted or undergoing gene therapy at the time of inclusion. Patients with graft failure without a new transplant may be included.

Exclusion Criteria:

* Carrier traits in autosomal recessive hereditary anemias

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients sustaining a confirmed or suspected diagnosis of an hereditary rare hemolytic anemia.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-11-13 (Actual); Primary Completion 2025-05-25 (Actual); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
To assess the prognostic value of LoRRca ektacytometry as biomarker providing information of SCD/RADs patients severity | Through study completion, an average of 2 year
  Severity was assesed as the occurence of:
  * Vaso-occlusive events (VOEs) in the last 24 months
  * Kidney injury (defined according to KDIGO guidelines)
  * Retinopathy (defined as proliferative and non proliferative)

SECONDARY OUTCOMES:
To investigate the correlation between LoRRca ektacytometry parameters and SCD/RADs patients genetic and phenotypic characterization. | Through study completion, an average of 2 year
  Genomic data will be generated using a targeted next-generation sequencing (tNGS) approach.
  Means, medians, standard deviations (SD), ranges and percentages were calculated using SPSS software (version 20, IBM SPSS Statistics, Chicago, IL, USA). Spearman's rank correlation was used to assess associations between variables. For comparing variables with two categories, either a student's t-test or a Mann-Whitney U test was performed, when appropriate. When the variable had more than two categories, an ANOVA or Kruskal Wallis test was used. A p value <0.05 was considered statistically significant.

CONTACTS AND LOCATIONS:
Locations (9):
- Spain (9):
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona
  - Hospital Sant Joan de Déu, Esplugues de Llobregat, Barcelona
  - Hospital General de Granollers, Granollers, Barcelona
  - Consorci Sanitari del Maresme - Hospital de Mataró, Mataró, Barcelona
  - Parc Taulí Hospital Universitari, Sabadell, Barcelona
  - Hospital Universitari Mútua de Terrassa, Terrassa, Barcelona
  - Consorci Sanitari de Terrassa, Terrassa, Barcelona
  - Hospital Universitari Arnau de Vilanova, Lleida, Lleida